CLINICAL TRIAL: NCT02958709
Title: Phase I/II Randomized, Open-label Trial to Evaluate the PK, Safety, and Outcomes of Treatment Including High Dose Rifampicin +/- Levofloxacin vs Standard Treatment for Pediatric Tuberculous Meningitis (TBM)
Brief Title: Optimizing Treatment to Improve TBM Outcomes in Children
Acronym: TBM-KIDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute for Research in Tuberculosis, Chennai, India (Unknown); University of North Carolina (Other); B. J. Medical College, Pune (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00051196; 1R01HD074944-01A1 (NIH)
Record Dates: First submitted 2016-09-13; First posted 2016-11-08 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2020-08

CONDITIONS: Tuberculosis, Meningeal
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Rifampin; Isoniazid; NSC 366140; Levofloxacin; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high dose RIF, INH, PZA, EMB (Experimental): Arm 1 participants will receive high-dose rifampicin for 8 weeks plus ethambutol at standard doses, in addition to standard doze pyrazinamide (PZA) and isoniazid.
  Interventions: Drug: High-dose: RIF, INH, PZA, EMB
- high dose RIF, INH, PZA, LEVO (Experimental): Arm 2 participants will receive high-dose rifampicin plus levofloxacin for 8 weeks, in addition to standard doze pyrazinamide and isoniazid.
  Interventions: Drug: High dose: RIF, INH, PZA, LEVO
- standard dose RIF, INH, PZA, EMB (Active Comparator): Arm 3 participants will receive standard of care dose rifampicin plus ethambutol for 8 weeks, in addition to standard doze pyrazinamide and isoniazid.
  Interventions: Drug: Standard of care: RIF, INH, PZA, EMB

INTERVENTIONS:
Drug: High-dose: RIF, INH, PZA, EMB — high-dose rifampicin plus standard dose H,Z,E, given for 8 weeks in treatment Arms 1 and 2
  Other Names: Rifampin
  Arms: high dose RIF, INH, PZA, EMB
Drug: High dose: RIF, INH, PZA, LEVO — high-dose rifampicin plus standard dose H,Z, with levofloxacin substituted for ethambutol for 8 weeks in treatment Arm 2
  Other Names: Levaquin
  Arms: high dose RIF, INH, PZA, LEVO
Drug: Standard of care: RIF, INH, PZA, EMB — standard doses of R,H,Z,E given for 8 weeks in treatment Arm 3, control arm.
  Other Names: control group
  Arms: standard dose RIF, INH, PZA, EMB

SUMMARY:
In this open-labeled, randomized clinical trial, the Investigator will assess the safety and pharmacokinetics (PK) of model-optimized doses of rifampicin (RIF) with or without levofloxacin (LEVO) given to children as part of multidrug treatment for tuberculous meningitis (TBM) versus standard treatment. The Investigators will also assess functional and neurocognitive outcomes by treatment group, as measured by the Pediatric Modified Rankin Score (MRS) and the Mullen Scales of Early Learning (MSEL), respectively.

DETAILED DESCRIPTION:
Open-label, randomized clinical trial in three treatment groups. Patients with probable or definite TB meningitis (TBM) will all receive isoniazid and pyrazinamide at standard doses for 8 weeks. Arm 1 participants will receive high-dose rifampicin plus ethambutol (EMB) at standard doses for 8 weeks. Arm 2 participants will receive high-dose rifampicin plus levofloxacin for 8 weeks. Arm 3 participants will receive rifampicin plus ethambutol at standard doses for 8 weeks (control arm). Patients will be screened to confirm TBM diagnosis, will receive 8 weeks of study treatment, and then will receive isoniazid (INH)/rifampicin for an additional 40 weeks, to complete 12 months of TBM treatment. All participants will receive oral steroids. PK sampling will be performed within first week and 6 (+/- 2) weeks following treatment initiation. Participants will have scheduled follow-up visits to assess safety and clinical status. In addition, functional and neurocognitive outcomes up to 18 months following treatment initiation will be assessed. Interim PK and safety analyses will be performed to ensure dosing is producing predefined PK targets and safety is acceptable. It is anticipated that a majority of children will be hospitalized for the initial 2-8 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 6kg
* Age ≥ 6 months to < 12 years and, in the opinion of the investigator, can tolerate the treatment and study participation.
* Probable or definite TBM according to diagnostic criteria or a positive Gene Xpert cerebrospinal fluid (CSF) test.
* Since participants will all be under legal age of independent consent, a parent or legal guardian must be willing and able to provide informed consent. If the subject is of appropriate age, she/he will also be asked to give assent if developmentally appropriate and clinically possible.
* Participant can comply with the protocol requirements in the opinion of the site investigator.

Exclusion Criteria:

* TB treatment for > 7 days
* Exposure via close contact with someone with multi drug resistant TB (MDR-TB) (or rifampicin mono-resistant TB) or personal history of MDR-TB (or rifampicin mono-resistant TB)
* Known intolerance or allergy to any of the study drugs
* Death imminent and expected within 24 hours, as assessed by the site investigator
* Moderate to severe renal or liver dysfunction (Grade 2 or higher abnormalities of creatinine, alanine aminotransferase (ALT), or direct bilirubin)
* HIV infection with any of the following:

Planned initiation of antiretroviral treatment (ART) during the experimental treatment phase (first 8 weeks), as initiation of ART is contraindicated in that time period with TBM.

On ART with planned continued use of a protease inhibitor or nevirapine (children can be switched to an acceptable alternative regimen and then participate)

* Having participated in other clinical studies with investigational agents or treatments within 8 weeks prior to enrollment.
* A clinically significant active medical condition or the presence of any concomitant severe illness or rapidly deteriorating health condition (outside of TB), which, in the opinion of the site investigator, would prevent appropriate participation in the trial, or that would make implementation of the protocol or interpretation of the study results difficult, or otherwise make the subject a poor candidate for a clinical trial.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Characterize the Volume of Distribution (Vd) in plasma of rifampicin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1-16
  Apparent volume of distribution estimated using population PK model
Characterize the Oral Clearance (CL/F) in plasma of rifampicin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1-16
  Examines the apparent total clearance of rifampicin from plasma after oral administration.
  Unit of Measure: Volume/time or volume/time/kg
Characterize the Rate of Absorption (ka) in plasma of rifampicin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1-16
  Examines the absorption rate constant for orally administered rifampicin. Unit of Measure: will be represented as a decimal.
Characterize the Penetration Coefficient in CSF of rifampicin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1 and 6
  Examines the ratio of CSF concentration to Plasma concentration of rifampicin Unit of Measure: will be represented as a decimal
Characterize the Volume of Distribution (Vd) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1-16
  Examines the apparent volume in which levofloxacin is distributed (i.e., the parameter relating drug concentration to drug amount in the body).
  Unit of measure: Liter (L)
Characterize the Volume of Distribution (Vd) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Week 4
  Examines the apparent volume in which levofloxacin is distributed (i.e., the parameter relating drug concentration to drug amount in the body).
  Unit of measure: Liter (L)
Characterize the Volume of Distribution (Vd) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Week 8
  Examines the apparent volume in which levofloxacin is distributed (i.e., the parameter relating drug concentration to drug amount in the body).
  Unit of measure: Liter (L)
Characterize the Volume of Distribution (Vd) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Week 16
  Examines the apparent volume in which levofloxacin is distributed (i.e., the parameter relating drug concentration to drug amount in the body).
  Unit of measure: Liter (L)
Characterize the Oral Clearance (CL/F) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1-16
  Examines the apparent total clearance of levofloxacin from plasma after oral administration.
  Unit of Measure: Volume/time or volume/time/kg
Characterize the Oral Clearance (CL/F) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Week 4
  Examines the apparent total clearance of levofloxacin from plasma after oral administration.
  Unit of Measure: Volume/time or volume/time/kg
Characterize the Oral Clearance (CL/F) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Week 8
  Examines the apparent total clearance of levofloxacin from plasma after oral administration.
  Unit of Measure: Volume/time or volume/time/kg
Characterize the Rate of Absorption (ka) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1-16
  Examines the absorption rate constant for orally administered levofloxacin. Unit of Measure: will be represented as a decimal.
Characterize the Rate of Absorption (ka) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Week 4
  Examines the absorption rate constant for orally administered levofloxacin. Unit of Measure: will be represented as a decimal.
Characterize the Rate of Absorption (ka) in plasma of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Week 16
  Examines the absorption rate constant for orally administered levofloxacin. Unit of Measure: will be represented as a decimal.
Characterize the Penetration Coefficient in CSF of levofloxacin given at model-derived optimal daily doses in children ages 6 months to 12 years of age with TBM. | Weeks 1 and 6
  Examines the ratio of CSF to Plasma concentration of levofloxacin Unit of Measure: will be represented as a decimal
Assess the relationship between RIF concentrations and longitudinal functional outcomes as measured by longitudinal Modified Rankin Score (MRS) for children | 48 weeks
  At the end of treatment, all participants' RIF concentrations (Cmax and AUC) will be compared across time against their MRS scores. MRS parameters and their scores (in parentheses) as follows: No symptoms at all (0),No significant disabilities despite symptoms in clinical examination; age appropriate behaviour and further development (1),Slight disability; unable to carry out all previous activities, but same independence as other age- and sex-matched children (no reduction of levels on the gross motor function scale) (2),Moderate disability; requiring some help, but able to walk without assistance; in younger patients adequate motor development despite mild functional impairment (reduction of one level on the gross motor function scale) (3), Moderately severe disability; unable to walk without assistance; in younger patients reduction of at least 2 levels on the gross motor function scale (4),Severe disability; bedridden, requiring constant nursing care and attention (5),
To evaluate the safety of TBM treatment over eight weeks, by treatment Arm, as measured by Grade 3 or higher adverse events | 8 weeks
  Grade 3 Adverse Events as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

SECONDARY OUTCOMES:
Describe neurocognitive outcomes among children ages 6 months to 6 years of age who are treated for TBM, longitudinally over 18 months, by treatmentArm, as measured by the Mullen Gross Motor Scale | 72 weeks
  The Gross Motor Scale is used to assess infants who are 33 months of age or younger and provides information about the child's kinesthetic experience.
  Maximum Raw Scores of Gross Motor Scale: 36 Raw scores are converted to T Scores (A type of standardized score) based on the child's age.
  A T Score has a mean of 50 and a standard deviation of 10. A T Score between 20 and 30 (or less than 20) has a descriptive category of "Very Low" A T Score between 31 and 39 has a descriptive category of "Below Average" A T Score between 40 and 60 has a descriptive category of "Average" A T Score between 61 and 69 has a descriptive category of "Above Average" A T Score between 70 and 80 has a descriptive category of "Very High"
Describe neurocognitive outcomes among children ages 6 months to 6 years of age who are treated for TBM, longitudinally over 18 months, by treatmentArm, as measured by the Mullen Visual Reception Scale | Week 72
  A cognitive score that may be derived from children ages birth to 68 months of age.
  The Visual Reception Scale assesses visual processing skills through isolation of oculomotor and visual-motor operations. This scale minimizes the motor output required to execute the response and eliminates the need for verbalized responses.
  Maximum Raw Scores of the Visual Reception Scale: 50 Raw scores are converted to T Scores (A type of standardized score) based on the child's age.
  A T Score has a mean of 50 and a standard deviation of 10. A T Score between 20 and 30 (or less than 20) has a descriptive category of "Very Low" A T Score between 31 and 39 has a descriptive category of "Below Average" A T Score between 40 and 60 has a descriptive category of "Average" A T Score between 61 and 69 has a descriptive category of "Above Average" A T Score between 70 and 80 has a descriptive category of "Very High"
Describe neurocognitive outcomes among children ages 6 months to 6 years of age who are treated for TBM, longitudinally over 18 months, by treatmentArm, as measured by the Mullen Fine Motor Scale | Week 72
  A cognitive score that may be derived from children ages birth to 68 months of age.
  The Fine Motor Scale emphasizes the output aspect of visual organization by assessing visual-motor skills, such as motor planning, motor control, and writing readiness.
  Maximum Raw Scores of the Fine Motor Scale: 49 Raw scores are converted to T Scores (A type of standardized score) based on the child's age.
  A T Score has a mean of 50 and a standard deviation of 10. A T Score between 20 and 30 (or less than 20) has a descriptive category of "Very Low" A T Score between 31 and 39 has a descriptive category of "Below Average" A T Score between 40 and 60 has a descriptive category of "Average" A T Score between 61 and 69 has a descriptive category of "Above Average" A T Score between 70 and 80 has a descriptive category of "Very High"
Describe neurocognitive outcomes among children ages 6 months to 6 years of age who are treated for TBM, longitudinally over 18 months, by treatmentArm, as measured by the Mullen Receptive Language Scale | Week 72
  A cognitive score that may be derived from children ages birth to 68 months of age.
  The Receptive Language Scale evaluates the ability to decode verbal input through tasks requiring auditory discrimination, linguistic conceptualization, sequencing, and use of spatial concepts.
  Maximum Raw Scores of the Fine Motor Scale: 48 Raw scores are converted to T Scores (A type of standardized score) based on the child's age.
  A T Score has a mean of 50 and a standard deviation of 10. A T Score between 20 and 30 (or less than 20) has a descriptive category of "Very Low" A T Score between 31 and 39 has a descriptive category of "Below Average" A T Score between 40 and 60 has a descriptive category of "Average" A T Score between 61 and 69 has a descriptive category of "Above Average" A T Score between 70 and 80 has a descriptive category of "Very High"
Describe neurocognitive outcomes among children ages 6 months to 6 years of age who are treated for TBM, longitudinally over 18 months, by treatmentArm, as measured by the Mullen Expressive Language Scale | Week 72
  A cognitive score that may be derived from children ages birth to 68 months of age.
  The Expressive Language Scale focuses on the child's use of spoken language for communication and expression during spontaneous utterances and during specific vocal or verbal responses to tasks.
  Maximum Raw Scores of the Fine Motor Scale: 50 Raw scores are converted to T Scores (A type of standardized score) based on the child's age.
  A T Score has a mean of 50 and a standard deviation of 10. A T Score between 20 and 30 (or less than 20) has a descriptive category of "Very Low" A T Score between 31 and 39 has a descriptive category of "Below Average" A T Score between 40 and 60 has a descriptive category of "Average" A T Score between 61 and 69 has a descriptive category of "Above Average" A T Score between 70 and 80 has a descriptive category of "Very High"
Describe TBM treatment outcomes at 12 months which will be classified as favorable (cured or treatment completed) or unfavorable (death, lost to follow up, treatment failure, transferred out) at 48 weeks. | 48 weeks
  TB treatment outcomes , favorable or unfavorable

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dooley, MD,PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- India (2):
  - Byramji Jeejeebhoy Government Medical College and Sassoon Hospital, Pune, Maharashtra
  - National Institute of Research in TB and Institute of Child Health, Chennai, Tamil Nadu
- UNC Project- Malawi, Lilongwe, Lilongwe District, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paradkar MS, Devaleenal D B, Mvalo T, Arenivas A, Thakur KT, Wolf L, Nimkar S, Inamdar S, Giridharan P, Selladurai E, Kinikar A, Valvi C, Khwaja S, Gadama D, Balaji S, Yadav Kattagoni K, Venkatesan M, Savic R, Swaminathan S, Gupta A, Gupte N, Mave V, Dooley KE; TuBerculous Meningitis in Kids (TBM-KIDS) Study Team. Randomized Clinical Trial of High-Dose Rifampicin With or Without Levofloxacin Versus Standard of Care for Pediatric Tuberculous Meningitis: The TBM-KIDS Trial. Clin Infect Dis. 2022 Oct 29;75(9):1594-1601. doi: 10.1093/cid/ciac208. PMID 35291004